CLINICAL TRIAL: NCT06961799
Title: Validating a Multifactorial Algorithm to Predict Fall Risk in Community Dwelling Older Persons Aged 65 Years or Older
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2024-0584
Record Dates: First submitted 2025-04-18; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Aged 65 Years or Older; Community Dwelling Older Adults; Falls Risk; Falls (Accidents) in Old Age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multifactorial algorithm to predict fall risk — In this new multifactorial algorithm we will add baseline data (personal characteristics, medical history, and physical and psychological measurements) to predict an older adults risk on falls. The accuracy of this new model will be tested with a 1-year follow up on falls.
  The new algorithm is inspired by the study of Lusardi et al. (2017): Lusardi MM, Fritz S, Middleton A, Allison L, Wingood M, Phillips E, Criss M, Verma S, Osborne J, Chui KK. Determining Risk of Falls in Community Dwelling Older Adults: A Systematic Review and Meta-analysis Using Posttest Probability. J Geriatr Phys Ther. 2017 Jan/Mar;40(1):1-36. doi: 10.1519/JPT.0000000000000099. PMID: 27537070; PMCID: PMC5158094.

SUMMARY:
Falls in older adults have an annual incidence between 23 and 34% for persons of 65 years and older. The lack of transfer of promising research results on falls prevention to daily practice may have several explanations. One of the first concerns for that matter may be a valid and sensitive selection of the persons at risk who are eligible for fall prevention interventions

Goals of the prospective obeservational study:

1. To validate a new, comprehensive, multifactorial screeningsintrument to predict the risk on falls in community dwelling, Belgian, older adults (>65years or older).
2. To optimize the new, comprehensive, multifactorial screeningsintrument and to specify correct cut off scores

Researchers will compare the data of the accuracy of new algorithm with the current Belgian policy.

Participants will participate in a one-time testing moment, where they will be asked some questions about general characteristics and medical history, followed by two questionnaire and seven physical tests . Based on this data, their fall risk will be assessed. In the year that follows, the older person's fall behavior will be monitored with a monthly falls calender. Participant will be asked to fill out these calenders everyday ('Did you fall today?' YES/NO) and send them at the end of each month to the researchers, digitally or postal.

DETAILED DESCRIPTION:
Two questionnaires:

1. Geriatric Depression Scale - 16
2. Falls Efficacy Scale - International

Seven physical tests:

1. Timed Up and Go
2. Times Up and Go with cognitive dual task (100 (repeatedly) minus 3)
3. Single Limb Stance
4. 5x Sit to Stand
5. 4meter Gait Speed
6. Tinetti
7. Four Balance Test

ELIGIBILITY:
Inclusion Criteria:

* 65years or older
* community dwellers
* absence of surgery or exacerbation of symptoms in the last 6 months
* ability to stand and walk independently (alone), possibly with an walking aid.

Exclusion Criteria:

* <65 years of age
* surgery within the previous 6 months affecting gait and mobility
* exacerbation of symptoms coming from a diagnosed disease
* older adults with insufficient (language) comprehension to complete the tests and questionnaires

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community dwelling, belgian older adults
Sampling Method: Non-Probability Sample
Enrollment: 228 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Conducted analysis of integraded tests | Baseline
  Fall risk calculated with the new multifactorial algorithm based on:
  * general, personal characteristics
  * medical history
  * physical measurements
  * self reported questionnaires
Number of falls among Belgian, community dwelling older adults | 1 year
  The number of falls measured with a monthly falls calender

SECONDARY OUTCOMES:
Depression | Baseline
  Measured with the Geriatric Depression Scale (GDS-16)
Fear of falling | Baseline
  Measured with the Falls Efficacy Scale (FES-I)
Functional mobility | Baseline
  Measured with the Timed Up and Go (seconds)
Executive cognitive capacity | Baseline
  Measured with the Timed Up and Go in combination with a cognitive dual task (100-3-3-3-...) (seconds)
Static Balance | Baseline
  Measured with the Single Leg stance (seconds)
Strength of the lower limbs | Baseline
  Measured with the 5x Sit to Stand (second)
Gait speed | Baseline
  Measured with the 4m Gait Speed (m/s)
Static and dynamic balance | Baseline
  Measured with the Tinetti: Performance-Oriented Mobility Assessment
Static Balance | Baseline
  Measured with the 4 balance test

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Cambier, Prof. Dr., Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium, Belgium